CLINICAL TRIAL: NCT03288259
Title: Transnasal Endoscopy in Obese Patients Are Candidates for Bariatric Surgery: Feasibility, Tolerance, Security and Cost-effectiveness.
Brief Title: Transnasal Endoscopy in Obese Patients Are Candidates for Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Amaury Teixeira Xavier, Principal Investigator, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 65003516.2.0000.5149
Record Dates: First submitted 2017-08-02; First posted 2017-09-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Transnasal endoscopy - Obesity - endoscopy without sedation
MeSH Terms: conditions — Obesity | interventions — Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese patients (Experimental): Obese patients undergoing Local Anesthetics and Transnasal Endoscopy.
  Interventions: Procedure: transnasal endoscopy; Drug: Local Anesthetics,Topical

INTERVENTIONS:
Procedure: transnasal endoscopy — Transnasal endoscopy without sedation with ultra-thin endoscopes in patients who are candidates for bariatric surgery
Drug: Local Anesthetics,Topical — Will be carried out topical anesthesia of the pharynx with lidocaine spray (10%) 6 puffs and instillation of nasal vasoconstrictor 4 drops.

SUMMARY:
Transnasal Endoscopy in Obese Patients are Candidates for Bariatric Surgery

Introduction and Objectives: high digestive endoscopy (HDE) is an important tool in the preoperative period of bariatric surgery. Patients with excess weight have a higher risk of cardiorespiratory complications during this procedure, being that the transnasal endoscopy (TNE) with an endoscope-thin is a safe alternative, comfortable and great value for money. The TNE allows the study of the upper gastrointestinal tract without the need for sedation. The objective of this work was to evaluate the feasibility, tolerance and safety of TNE in obese patients are candidates for bariatric surgery. Methods: This was a prospective study with all patients with indication for surgery of obesity undergoing endoscopic transnasal preoperatively, between December 2016 and August 2018, at the Hospital of the Federal University of Minas Gerais. The variables evaluated were: age, gender, suitability of the exam, tolerance by the patient through the visual analogue scale, incidence of complications and need for sedation. Oxygen saturation, heart rate and systolic blood pressure were recorded. Conclusion: The transnasal endoscopy is a feasible alternative, well tolerated and safe the conventional endoscopy in evolution the preoperative bariatric surgery. The benefits of transnasal endoscopy in obese patients mainly consist in carrying out the procedure without sedation, which may provide reduction of risks, costs and waive the need for a companion. Key words: transnasal endoscopy - Obesity - endoscopy without sedation.

DETAILED DESCRIPTION:
1. - Introduction - scientific background, relevance and rationale of the research

   According to data from 2014 of the World Health Organization (WHO), globally there are more than 1.9 billion adults are overweight and at least 600 million obese. 39% of adults above 18 years were overweight and 13% were obese that year. According to the WHO classification, the population with overweight is one that has a body mass index (BMI) greater than or equal to 25 kg/m² and has a BMI greater than or equal to 30 Kg/m² is obese.

   In Brazil, the excess weight also assumes epidemic proportions. The most recent survey of the Ministry of Health (MH) conducted in 2014 found that more than half of the Brazilian population is overweight (52.5%) and of these, 17.9% are obese. The prevalence of obesity has doubled during the period between 1980 and 2014 in Brazil. The data are disclosed annually by MH since 2006. Obesity and overweight are considered risk factors relevant to chronic diseases such as diabetes mellitus type 2, cardiovascular diseases and malignant neoplasms.

   Among the various treatment modalities, the bariatric surgery is an effective remedy in cases of morbid obesity with a failure of clinical treatment, giving patients a reduction of mortality rates and resolution of clinical comorbidities, as was demonstrated in an observational study of ten years of follow-up.

   The reason for indication of high digestive endoscopy (HDE) in the pre-operative bariatric surgery refers to the detection and/or treatment of injuries that could affect the type of proposed surgery, causing complications in the immediate postoperative period or result in symptoms after surgery. However, the endoscopic examination of routine pre-operative in these patients is controversial if there is no gastrointestinal symptoms studies. One of the reasons for this, concerns the increased cardiovascular risk of obese subjects associated with sedation. In Brazil as well as in other centers, the guidelines recommend HDE with research of Helicobacter pylori infection in all patients preoperatively of bariatric surgery. The traditional HDE involves the use of conscious sedation, with a mortality rate of 0.03% and morbidity of 0.54%. Adverse cardiopulmonary related to sedation and analgesia equivalent to about 60% of the complications of high digestive endoscopy, and such complications are more frequent in obese patients.

   It is important to highlight the high prevalence of obstructive sleep apnea (OSA) in morbidly obese patients, some studies suggest up to 68%. The OSA is a syndrome characterized by periods of partial or complete obstruction during sleep, which is more common in obese individuals. OSA may cause hypoxemia, hypercarbia and cardiovascular dysfunction. BMI > 30 kg/m² is a risk factor known for hypoxemia in subjects undergoing endoscopic procedures. Small doses of opioids and benzodiazepines may cause deep sedation and obstruction of the airway is high in obese patients who have obstructive sleep apnea.

   The endoscopy by transnasal (TNE), founded in 1994, uses ultrathin endoscopic from 5 to 6 mm in diameter that can be introduced through the nasal passages allowing complete study of upper gastrointestinal tract including the possibility of realization of biopsies and other small interventions. The main advantage of the TNE is to dispense with the use of sedation, making the endoscopic procedure safer for patients who have cardiorespiratory risk and anesthesia higher. Moreover, compared to conventional HDE the costs involved in the TNE are significantly lower.

   Few studies have compared the TNE with conventional HDE. A Japanese study measured the diagnostic efficacy of the TNE compared to HDE. This study found that the resolution of images endoscopy was similar between the two modalities. Sensitivity, specificity and accuracy of transnasal were 90, 100 and 93%, respectively. One of the largest series evaluated 1100 patients undergoing TNE, with satisfactory results in 94% of patients. In the same study, 91% of patients who had undergone prior to conventional endoscopy preferred the transnasal. A multicenter study published in 2003 showed a significant difference in cost between the HDE and the TNE. The average total cost of the procedure was 512 US dollars (+/- 100.8 US dollars) for HDE with sedation and 328.6 US DOLLARS (+/- 70.3 US dollars) for TNE without sedation (p<0.0001).

   After extensive research in major databases of literature, the investigators found only one study that examined the use of the TNE in obese patients are candidates for bariatric surgery. In this study, Nigeria Tome et al., 25 patients were allocated. The variables analyzed were suitability of examination, patient tolerance, need for sedation and ability to carry out interventions. Significant pathological alterations during the endoscopic examination were present in 14 patients (56%), which included hiatal hernia (28%), gastritis (16%), intestinal metaplasia in the esophagus (12%), gastric polyps (8%), gastric ulcer (4%) and varices (4%). In all participants reached the second duodenal portion with excellent tolerance. There was no need for sedation in 23 patients (92%). biopsies were indicated in 12 participants and successful in all 12 (100%).

   The TNE has been validated, mainly in Japan, for screening of gastric cancer early. Although the TNE is still little used in the west, is considered an attractive alternative for patients with cardiovascular comorbidities and important respiratory the example of elderly and obese. Since 2009, our center has developed lines of research related to the use of the TNE in specific populations, such as for screening of esophageal neoplasm in high risk patients and for the screening of esophageal varices in end-stage cirrhosis. In the literature, there is no publication concerning the use of the TNE in obese patients in Brazil and Latin America.
2. - The research objectives

   This prospective clinical study, has the objective of evaluating the feasibility, the acceptance of the patient, the safety and the costs involved using the TNE in obese patients are candidates for bariatric surgery.
3. - Materials and Methods

   Design:

   Prospective study proposed to be initiated after approval by The Ethics Committee and completed by August 2018. The target of the study of approximately 100 patients, based on the expectation of new cases per month of patients who are candidates for bariatric surgery the outpatient obesity. The demand of the ambulatory of Digestive System Surgery of the Clinicals Hospital of Minas Gerais is on average of 5 new cases per month.

   Inclusion criteria:

   Patients referred to the endoscopy of the Institute Alfa of Gastroenterology of the Clinicals Hospital (IAG-HCUFMG) by the Digestive System Surgery and which meet the following criteria:

   Between the ages of 18 and 65 years. A BMI greater than or equal to 40 Kg/m² or greater or equal 35 Kg/m² associated with comorbidity; The absence of contraindications to bariatric surgery; Voluntary acceptance to be submitted to the transnasal endoscopy; Agreed to participate in the study and sign the informed consent form (ICF).

   Exclusion criteria:

   Surgery, fractures or nasal malformations in advance; History of epistaxis; Allergy to components of the topical anesthetic used prior to the examination; Coagulation disorders or use of anticoagulants; Pregnancy; Psychiatric disorder important; Clinical contraindication to the examination of high digestive endoscopy;

   Procedure:

   The procedure of transnasal endoscopy will be performed by endoscopists trained in the technique, industry members of Gastrointestinal Endoscopy of the IAG-HCUFMG. The information from the questionnaires will be collected by members of the service. The ultra-thin endoscope with a diameter of 5.9 mm and working channel of 2 mm, with digital chromoscopic, will be used in exams. The representative images of the examination will be recorded and photographed. The patients will be monitored with pulse oximetry and ECG monitor for assessment of heart rate, blood pressure and oxygen saturation. If necessary, will be provided supplemental oxygen via nasal catheter.

   Before the TNE, will be carried out topical anesthesia of the pharynx with lidocaine spray (10%) 6 jets and instillation of nasal vasoconstrictor. The procedures initially will be performed without sedation. However if the degree of discomfort is high, or nasal cavity does not allow the passage of the endoscope, can be used to oral administration, at the discretion of the endoscopist.

   The exam will be considered complete if the appliance reaches the second duodenal portion and is performed retroflex, allowing the visualization of all portions of the digestive system and the achievement of biopsies if necessary. The samples of biopsies will be obtained by collet pediatric 1.8 mm.

   The tolerance of the patient will be assessed through a visual analogue scale (VAS) from 0 to 10 (0 - no discomfort; 10 - unbearable) which will be completed by the patient after the examination, at the request of an independent researcher. Another parameter to measure the level of comfort of the patient will be performed by the physician endoscopist wizard, who uses VAS to efforts of vomiting and intolerance, being 0 for no reflection of vomiting and 10 to violent efforts.

   The safety of the procedure of TNE will be evaluated by the rate of complications and side effects that occurred (cardiorespiratory impairment, epistaxis, nasal pain, reaction vessel vagal-) and by the index called double product (DP). The heart rate (HR), blood pressure and oxygen saturation will be documented before, during and after the procedure. The double product will be the product of the systolic blood pressure and heart rate (SBP X HR). The DP reflects the myocardial oxygen consumption and cardiac output in tests of effort, being a tool the prognosis of mortality in cardiac patients during rest and exercise. A value greater than 15000 is indicative of cardiovascular stress considerably. The cardiovascular stress serves to evaluate both the safety of the procedure as well as the comfort of the patient according to the literature.

   Shall be assessed the cost of the TNE compared with the conventional HDE. To do this will be compared the values of inputs, materials and medicines needed. The researchers will use as the basis for these calculations the updated values of medicinal products and inputs used during sedation. Will be considered the table of the Unified Health System (SUS) as the main reference. There will be a real comparison of costs between the two methods of examination. For this reason, will be calculated the values of medicinal products and inputs used in 100 patients undergoing traditional endoscopy comparing costs with the group of candidates in the study that pass through the transnasal endoscopy. Similar profiles of patients will be allocated and the same researchers conduct the tests in both groups and at the same institution.

   All patients will complete a questionnaire 15 to 30 minutes after the transnasal endoscopy and will be released next to the house.

   Collected Data and Statistical Analysis:

   Will be collected general data of patients such as age, gender, BMI, comorbidities, medications in use, history of allergic reactions, type of bariatric surgery proposal, history of previous surgeries, previous experience with endoscopic procedures and vital data. On the exam will be collected information about the endoscopic findings, biopsies, complications and adverse reactions, patient tolerance and expenses. After the procedure, the degree of patient satisfaction will also be analyzed in questionnaire.

   All of this information and the results will be compared with the main data in the literature. Bivariate analyzes shall be calculated from the test "t" test for continuous variables and the chi-square test or Fisher exact test for categorical variables. Proportions will be reported by categorical data; and mean, median and standard deviation for continuous variables. P values less than 0.05 are considered statistically significant.
4. - Plan for the collection and analysis of data

   The study will be conducted as schedule shown below:

   Collection of cases - After approval by The Ethics Committee Literature Survey - 12/2015 to 12/2017 Preliminary analysis of the results - 12/2017 Final analysis of results - 12/2017 to 06/2018 Copyrighting - 12/2017 to 08/2018 Presentation - 08/2018
5. - critical analysis of the potential risks and benefits

   The patients will be submitted to the transnasal endoscopy and biopsies as a way of assessing the upper gastrointestinal tract in the pre-operative bariatric surgery. It is a procedure mandatory before surgery for obesity. The risks related to the endoscopic procedure are very low. The TNE will be performed by experienced endoscopists of clinical staff of the Clinicals Hospital and in an environment that has all the human and material resources for hemodynamic monitoring and cardiopulmonary resuscitation.

   The main complications as the endoscopic procedure are: epistaxis, nasal pain, gastrointestinal bleeding, perforation, infection, need for surgery, sepsis and death. To minimize the risks, the hospital offers equipment for basic and advanced life support in addition to trained personnel in these situations The benefits of transnasal endoscopy in this group of patients (obese) consist primarily in performing the procedure without sedation, which may provide reduction of risks, costs and waive the need for a companion.
6. - Plan for dissemination of results

   The results of this study will be presented at conferences and published in specialized journals of recognized credibility. These results will compose the masters thesis to be defended by the Graduate Program in Applied Sciences to Adult Health, concentration area in Applied Sciences the digestive tract.
7. - explanation of the criteria to stop or suspend the search

   After the beginning of the collection of cases, if this happens to any complications or unexpected deaths, the work will be suspended immediately or even stopped on duty, and the Committee on Ethics statement without holding.
8. - Place of Research

   The survey will be conducted in the upper digestive endoscopy of the Institute Alfa of Gastroenterology at the Clinicals Hospital of UFMG.
9. - Budget detailed financial

The resources for completion of endoscopic procedure and histopathological diagnosis, expenditures on inputs, drugs and human material are already part of the list of procedures covered by SUS. There is no additional cost to the institution or to the patient. Therefore, this study will not charge for the Clinicals Hospital, as financial resources are already covered by the Public Health System and the procedure is already part of the routine of the Digestive Endoscopy of the Institute Alfa of Gastroenterology.

ELIGIBILITY:
Inclusion Criteria:

* A BMI greater than or equal to 40 Kg/m²
* A BMI greater or equal 35 Kg/m² associated with comorbidity (e.g., arterial hypertension, diabetes, dyslipidemia, sleep apnea)

Exclusion Criteria:

* Surgery, fractures or nasal malformations
* History of epistaxis
* Allergy to components of the topical anesthetic used prior to the examination
* Coagulation disorders or use of anticoagulants
* Pregnancy
* Psychiatric disorder important

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the procedure | 15 minutes
  The exam will be considered feasible if the appliance reaches the second duodenal portion and is performed retroflexão, allowing the visualization of all portions of the digestive system and the achievement of biopsies if necessary.
  All patients will complete a questionnaire 15 to 30 minutes after the transnasal endoscopy and will be released next to the house.
  All of this information and the results will be compared with the main data in the literature. Bivariate analyzes shall be calculated from the test "t" test for continuous variables and the chi-square test or Fisher exact test for categorical variables. Proportions will be reported by categorical data; and mean, median and standard deviation for continuous variables. P values less than 0.05 are considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Alpha Institute of Gastroenterology - HC/UFMG Rua Alfredo Balena, 110 - 2. Cycling - Santa Efigênia., Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
Participants can be identified by the number of medical records and phone contacts have been duly authorized by the institution responsible.